CLINICAL TRIAL: NCT02560285
Title: An International Multicenter Prospective Study for Identify High-risk Patients in Cardiac Surgery Procedures: HiriSCORE
Brief Title: High-risk Patients in Cardiac Surgery Procedures: HiriSCORE
Acronym: HiriSCORE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: InCor Heart Institute (Other); Cardiology Institute of the Distrito Federal, Brazil (Unknown); Clinical Hospital Samuel Libânio of Pouso Alegre, Brazil (Unknown); Beneficência Portuguesa de São Paulo (Other); National Institute of Cardiology, Laranjeiras, Brazil (Other Government); Russian Cardiology Research and Production Center, Russia (Unknown); Chinese Academy of Medical Sciences, Fuwai Hospital (Other); TotalCor Hospital, Brazil (Unknown); Dante Pazzanese Institute of Cardiology, Brazil (Unknown); Santa Casa de Misericórdia of Marília, Brazil (Unknown); Hospital de Base (Other); Novosibirsk Cardiology Recearch and Production Center, Russia (Unknown)
Responsible Party: Sponsor
Other Study IDs: USaoPauloGH1001; 1.289.986 (Other: Ethics Committee for the Analysis of Research Projects)
Record Dates: First submitted 2015-06-30; First posted 2015-09-25 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-10

CONDITIONS: C.Surgical Procedure; Cardiac
Keywords: Risk assessment; Mortality; Morbidity; Risk factor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Development / 2000 participants: * Age >18 years;
  * Patients undergoing cardiac surgery procedures (elective, urgent or emergency) for CABG; heart valve surgery; CABG + heart valve surgery; ascending aorta surgery + heart valve surgery or CABG, who have mortality risk with STS score>5 or EuroSCORE II>5.
- Validation / 1000 participants: * Age >18 years;
  * Patients undergoing cardiac surgery procedures (elective, urgent or emergency) for CABG; heart valve surgery; CABG + heart valve surgery; ascending aorta surgery + heart valve surgery or CABG, who have mortality risk with STS score>5 or EuroSCORE II>5.

SUMMARY:
Over time there is a need to improve old and develop new risk models. Overall the assessment of mortality risk in cardiac surgery is performed with the use of preoperative risk models. The use of improved risk models and increased accuracy in the technique of preparing these mathematical systems does not have a positive impact on the level of prediction, which is still inaccurate, especially in the considered group of high risk. New models need to be built not only for a better prediction of mortality risk, if not also to predict morbidity in the group of patients at higher risk of complications after cardiac surgery procedures.

The aim of this study is:

* To construct the HiriSCORE to identify patients at higher risk of complications after cardiac surgery procedures
* Assessing the impact of pre-, intra- and postoperative period to the prognosis of morbidity and mortality in high-risk patients undergoing cardiac surgery procedures.

DETAILED DESCRIPTION:
The risk predicts models are the mathematical tools for identification of the patients with complications risk after cardiac surgery procedures.

Over time, however, due to technical progress (the development of hybrid surgery, new valves and prostheses), the development of new drugs, changes in the environment and social conditions in which do patients live, there is a need to improve old and develop new models. Based on the statement that high risk patients have similar characteristics (clinical and laboratory) regardless of the procedure to which they were submitted, creating a new risk score to this group of patients must be sought. Improving the model quality was achieved by using more accurate risk assessments. In general, the assessment of mortality risk in cardiac surgery is performed with the use of preoperative risk models (EuroSCORE II, STS-score). However, the use of improved risk models and increased accuracy in the technique of preparing these mathematical systems, unfortunately, does not have a positive impact on the level of prediction, which is still inaccurate, especially in the considered group of high risk. New models need to be built not only for a better prediction of mortality risk, if not also to predict morbidity in the group of patients at higher risk of complications after cardiac surgery procedures.

The aim of this study is:

* To construct the HiriSCORE to identify patients at higher risk of complications after cardiac surgery procedures (the investigators have proposed a high-risk evaluation criteria: EuroSCORE II> 5 or STS-score> 5);
* Assessing the impact of pre-, intra- and postoperative period to the prognosis of subsequent morbidity and mortality in high-risk patients who have passed cardiac surgery procedures.

It was decided to conduct this research in two phases. The developmental phase is carried out for 30 months and includes an analysis of at least 2,000 patients who will pass cardiac surgery procedures in institutions and hospitals involved in the study. After this analysis, including outcomes, will be constructed the HiriSCORE, a new test-model for high-risk patients. In the validation phase of the study, which will involve a further 1,000 patients it is planned preparation and verification of effectiveness of the HiriSCORE model where it will be compared to the STS Score and the EuroSCORE II.

The study will include the patients of 18 years old or older who have undergone cardiac surgery procedures, such as coronary artery bypass grafting (isolated or combined with any heart valve intervention), heart valve surgery, and surgery on the ascending aorta (only combined with operations on the aortic valve or CABG).

Totally, it is proposed assessment of 170 variables (factors perceived risk) for each patient (preoperative, intraoperative, and up to 12 hours after surgery).

The study of mortality and postoperative complications such as renal replacement therapy, stroke, reoperation for bleeding, respiratory failure, cardiogenic shock, will be carried out within 30 days after cardiac surgery procedures.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing cardiac surgery procedures, such as coronary artery bypass grafting, heart valve surgeries, co-operations on aorta and valve or CABG and variations of this procedures, regardless of the operation or treatment outcomes
* Mortality risk with STS score>5 or EuroSCORE II>5

Exclusion Criteria:

* Isolated surgery on ascending aorta, aortic arch or descending aorta
* Heart transplantation
* Impossibility to include patient´s data in research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing cardiac surgery procedures
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2016-01 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
Mortality analysis | 30 days
  Patient´s mortality data collection following 30 days after the main procedure

SECONDARY OUTCOMES:
Stroke with neurological consequences (pareses or plegia) | 30 days
  Stroke with neurological consequences (pareses or plegia) following 30 days after the main procedure
ST-elevation Myocardial infarction | 30 days
  ST- elevation Myocardial infarction following 30 days after the main procedure
Non- ST- elevation Myocardial infarction | 30 days
  Non- ST- elevation Myocardial infarction following 30 days after the main procedure
Deep sternal wound infection | 30 days
  Deep sternal wound infection following 30 days after the main procedure
Bleeding requiring reoperation | 30 days
  Bleeding requiring reoperation following 30 days after the main procedure
Sepsis | 30 days
  Sepsis following 30 days after the main procedure
Endocarditis | 30 days
  Endocarditis following 30 days after the main procedure
Respiratory failure | 30 days
  Respiratory failure following 30 days after the main procedure
Renal replacement therapy | 30 days
  Renal replacement therapy following 30 days after the main procedure
Hepatic failure | 30 days
  Hepatic failure following 30 days after the main procedure
Unplanned cardiac reoperation | 30 days
  Unplanned cardiac reoperation following 30 days after the main procedure
Unplanned cardiac percutaneous intervention | 30 days
  Unplanned cardiac percutaneous intervention following 30 days after the main procedure

CONTACTS AND LOCATIONS:
Overall Officials: Fábio B Jatene, MD, PhD, Study Chair — Heart Institute of São Paulo Medical School; Omar AV Mejía, MD, PhD, Study Director — Heart Institute of São Paulo Medical School; Maxim D Goncharov, MD, Principal Investigator — Heart Institute of São Paulo Medical School; Camila PS Arthur, MD, Principal Investigator — Heart Institute of São Paulo Medical School; Ricardo R Dias, MD, PhD, Principal Investigator — Heart Institute of São Paulo Medical School; Carlos MA Brandão, MD, PhD, Principal Investigator — Heart Institute of São Paulo Medical School; Rodrigo C Segalote, MD, Principal Investigator — National Cardiology Institute; Diego M Ferreira, MD, Principal Investigator — National Cardiology Institute; Marcos G Tiveron, MD, PhD, Principal Investigator — Santa Casa de Misericórdia of Marília; Helton A Bomfim, N, Principal Investigator — Santa Casa de Misericórdia of Marília; Renat Suleimanovich Akchurin, MD, PhD, Principal Investigator — Russian Cardiology Research and Production Center; Elina Evgenievna Vlasova, MD, Principal Investigator — Russian Cardiology Research and Production Center; Pedro Gabriel M de Barros e Silva, MD, PhD, Principal Investigator — TotalCor Hospital; João Galantier, MD, Principal Investigator — TotalCor Hospital; Alexandre C Hueb, MD,PhD, Principal Investigator — Clinical Hospital Samuel Libânio of Pouso Alegre; Maurício LJ Guerrieri, MD, Principal Investigator — Clinical Hospital Samuel Libânio of Pouso Alegre; Marcelo A Nakazone, MD, PhD, Principal Investigator — Hospital de Base of São José de Rio Preto; Mauricio N Machado, MD, PhD, Principal Investigator — Hospital de Base of São José de Rio Preto; Fernando A Atik, MD, PhD, Principal Investigator — Cardiology Institute of the Distrito Federal; Murilo T Macedo, MD, Principal Investigator — Cardiology Institute of the Distrito Federal; Luís RP Dallan, MD, Principal Investigator — Heart Institute of São Paulo Medical School; José AD Santiago, MD, Principal Investigator — Heart Institute of São Paulo Medical School; Elinthon T Veronese, MD, Principal Investigator — Heart Institute of São Paulo Medical School; Pablo MA Pomerantzeff, MD, PhD, Principal Investigator — Heart Institute of São Paulo Medical School; Luiz Augusto F Lisboa, MD, PhD, Principal Investigator — Heart Institute of São Paulo Medical School; Luís Alberto O Dallan, MD, PhD, Principal Investigator — Heart Institute of São Paulo Medical School; Shengshou Hu, MD, PhD, Principal Investigator — Fuwai Hospital and Cardiovascular Institute; Zhe Zheng, MD, PhD, Principal Investigator — Fuwai Hospital and Cardiovascular Institute; Heng Zhang, MD, PhD, Principal Investigator — Fuwai Hospital and Cardiovascular Institute; Alexander Bogachev-Prokofiev, MD, PhD, Principal Investigator — Novosibirsk Cardiology Recearch and Production Complex; Magaly Arrais dos Santos, MD, PhD, Principal Investigator — Instituto Dante Pazzanese de Cardiologia; Jenny Rivas de Oliveira, MD, Principal Investigator — Instituto Dante Pazzanese de Cardiologia; Luiz C Bento de Souza, MD, PhD, Principal Investigator — Instituto Dante Pazzanese de Cardiologia; Jóse H Palma da Fonseca, MD, PhD, Principal Investigator — Heart Institute of São Paulo Medical School; Filomena Regina BG Galas, MD, PhD, Principal Investigator — Heart Institute of São Paulo Medical School; Ludhmila A Hajjar, MD, PhD, Principal Investigator — Heart Institute of São Paulo Medical School; Roberto Kalil Filho, MD, PhD, Principal Investigator — Heart Institute of São Paulo Medical School
Locations (1):
- Fabio B Jatene, MD, PhD, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
All data can be used by centers coparticipants after approval by the HiriSCORE group.